CLINICAL TRIAL: NCT02933957
Title: Chinese Arteriosclerosis Series Evaluation-She Minority Study
Acronym: CASE-SMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Shougang Hospital (Other)
Collaborators: MinDong Hospital of Ningde City (Unknown)
Responsible Party: Principal Investigator, Hongyu Wang, Director and Professor of Vascular Medicine, Peking University Shougang Hospital
Other Study IDs: PUShougangH
Record Dates: First submitted 2016-10-08; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Vascular Disease
Keywords: Vascular Evaluation; influencing factor; She Minority population
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Traditionally, people have always been focusing on vascular injuries by angiography. Recent years, the investigators have further known that the pathological foundation of various cardiovascular complications not only lies in the vascular lumen, but also vessel wall. Therefore, now it is possible to detect and prevent vascular disease early. There are many influencing factors on functional and structural damages of vessels, including genetic and environmental factors. The investigators have done many researches on populations of the Han nationality, which has the largest population in China. Thus, the investigators further wonder whether the function and structure of vessel differ in the She Minority of a remote southern region in China. The investigators will enroll 150 subjects of two ethnic groups respectively in the local population， namely She Minority and Han nationality. All subjects enrolled into the study will complete a questionnaire survey of the general situation and conduct vascular related examinations, including evaluation of arterial stiffness, arterial elasticity indexes, subclinical carotid atherosclerosis and biomarkers. The investigators will analysis vascular differences between the two populations and provide a theoretical basis for the specific strategies of prevention and treatment.

DETAILED DESCRIPTION:
Population Subjects volunteered to participate the study will be all enrolled into the study. The study is designed to enroll subjects from two ethnic groups in the local population, namely She Minority and Han nationality. All participants will be asked to sign a written informed consent and the study has been approved by the hospital.

Methods

1. Questionnaire The questionnaire survey included family history, disease history (including coronary artery disease, cerebrovascular disease, hypertension, diabetes mellitus, peripheral artery disease), medication history (including cardiovascular drugs, hypertension drugs, diabetes drugs, lipid-lowering drugs), physical activity, smoking condition, drinking status, dietary and life habits etc.
2. Arterial stiffness by vascular function apparatus Arterial stiffness is assessed by brachial-ankle pulse wave velocity (ba-PWV) using an automatic vascular function apparatus. Subjects lie on the detection bed resting about 10 minutes and the apparatus record the value of ba-PWV automatically.
3. Peripheral artery detection by vascular function apparatus Ankle-brachial index (ABI) is used as an evaluation index of peripheral artery and can be measured by an automatic vascular function apparatus.

   During the detection of ABI, the blood pressure of the four limbs will be measured simultaneously.
4. Arterial elasticity indexes by carotid ultrasound apparatus A Doppler ultrasound apparatus with a built-in software named quality arterial stiffness (QAS) will be used to measure arterial elasticity indexes, including stiffness coefficient β, pressure strain elastic coefficient, arterial compliance etc.
5. Subclinical carotid atherosclerosis by carotid ultrasound apparatus Assessment indexes of subclinical atherosclerosis including carotid intima-media thickness (IMT), carotid plaque, carotid internal diameter， carotid blood flow peak velocity, diastolic peak velocity of carotid artery, average velocity, resistance index (RI) and pulsation index (PI) will be measured by Doppler ultrasound apparatus.

   A more qualified detection of IMT will be also complete by a Doppler ultrasound apparatus with a built-in software named quality intima-media thickness (QIMT).
6. Vascular endothelial function detection Vascular endothelial function will be assessed by a noninvasive method of brachial ultrasound, named flow mediated dilation (FMD). Subjects lie on the detection bed resting 10 minutes and the operator will detect two times of the brachial artery diameter before and after hyperemia.
7. Biomarkers Biomarkers including fasting plasma glucose, plasma lipids (including total cholesterol, triglyceride, low density lipoprotein cholesterol, high density lipoprotein cholesterol), blood uric acid, blood urea nitrogen, creatinine, high sensitive C reactive protein, homocysteine lipoprotein a, Apolipoprotein A1, Apolipoprotein B, glycosylated hemoglobin, insulin, C-peptide etc.

Statistical analysis The investigators will take the double input and check all data. Statistical Product and Service Solutions (SPSS Version 20.0 ) will be the software of analyzing.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are natural population, from She Minority in Fujian province
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
value of brachial ankle pulse wave velocity | one and a half years

SECONDARY OUTCOMES:
Percentage of flow mediated dilation | one and a half years
Value of arterial elasticity including stiffness coefficient β, pressure strain elastic coefficient, arterial compliance | one and a half years
Thickness of carotid intima-media by carotid ultrasound | one and a half years
  Carotid ultrasound will be used to measure the thickness of carotid intimate-media.
Presence of Carotid Plaque | one and a half years
  Carotid ultrasound will be used to measure the presence of carotid plaque according to Mannheim Consensus
Number of peripheral arteriosclerosis occlusion measured by ankle brachial index | one and a half years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Shougang Hospital, Beijing, Beijing Municipality, China